CLINICAL TRIAL: NCT06746948
Title: Prevalence and Influencing Factors of the Dyadic Psychological Stress Among Patients With Lung Cancer and Their Family Caregivers: A Cross-Sectional Study
Brief Title: Dyadic Psychological Stress Among Lung Cancer Patient-caregiver Dyads
Status: Completed | Type: Observational
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Juan LI, lecturer, Central South University
Other Study IDs: Dyadic psychological stress
Record Dates: First submitted 2024-12-15; First posted 2024-12-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancers; Lung Cancer Patients
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lung cancer caregiver-caregiver dyads
  Interventions: Other: dyadic psychological distress

INTERVENTIONS:
Other: dyadic psychological distress — There is no intervention among the cross-sectional study.

SUMMARY:
A lung cancer diagnosis has a huge impact on the psychological well-being of both patients and family caregivers. However, the current psychological stress status among dyads remains unclear. The investigators aimed to determine the prevalence of anxiety and depression and identify the factors that influence patients with lung cancer and their caregivers. The investigators will conduct a cross-sectional study of 254 dyads of lung cancer patients and family caregivers from four tertiary hospitals in Hunan Province, China from January 2021 to June 2021. Besides, the investigators used several instruments to collect data on depression, anxiety, illness perception, mindfulness, self-compassion, and dyadic coping. The independent samples t-test, analysis of one-way variance, Spearman's correlation analysis, and multiple linear regression analysis were employed. The results will recommend oncology nurses promptly screen high-risk patient-caregiver dyads who may suffer from severe psychological stress and provide them with targeted psychosocial interventions.

ELIGIBILITY:
Inclusion Criteria:

* As for patients: aged≥18 years; hospitalized patients with lung cancer diagnosed by pathological section or cytology; and relatively stable condition, conscious, and able to express their willingness correctly.
* As for caregivers: aged ≥18 years; a primary caregiver with a cumulative caregiving time of more than 33 hours; and a family member of the patient with lung cancer, such as spouse, children, parents, or other relatives.

Exclusion Criteria:

* As for patients: people with a combination of other cancers or serious life-threatening diseases; the presence of audiological disorders or previous mental or cognitive disorders, such as anxiety disorder, or depression disorder; and receiving mental disorder treatments.
* As for caregivers: formal caregivers with employment relationships, such as nannies; the presence of audiological disorders or previous mental disorders or cognitive disorders, such as anxiety disorder, depression disorder; and receiving mental disorder treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized patients with lung cancer diagnosed by pathological section or cytology and a primary caregiver with a cumulative caregiving time of more than 33 hours; and a family member of the patient with lung cancer, such as spouse, children, parents, or other relatives.
Sampling Method: Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
depression | From enrollment through study completion, an average of 6 months
  The investigators measured dyadic depressive symptoms using the Patient Health Questionnaire-9 (PHQ-9), which is a 9-item questionnaire. Scores range from 0 to 27, with higher scores indicating more severe depression. According to Kroenke et al.'s scoring of the PHQ-9, a score of 0-4 indicates no depression, 5-9 indicates mild depression, 10-14 indicates moderate depression, 15-19 indicates moderate severe depression, and 20-27 indicates severe depression. The prevalence of depression is equal to the number of cases with a PHQ-9 score of 5 or greater divided by the total number of cases. Cronbach's alpha coefficients in this study were 0.85 and the KMO test value was 0.719, which showed good reliability and validity.
anxiety | From enrollment through study completion, an average of 6 months
  The investigators assessed anxious symptoms using the Generalized Anxiety Disorder-7 scale (GAD-7), which is a 7-item questionnaire. Scores range from 0 to 21, with higher scores indicating more severe anxiety. According to Spitzer et al's evaluation of GAD-7 scale, a score of 0-4 indicates no anxiety, 5-9 indicates mild anxiety, 10-14 indicates moderate anxiety, and 15-21 indicates severe anxiety. The prevalence of anxiety was defined as the number of cases with a GAD-7 score of 5 or greater divided by the total number of cases. Cronbach's alpha coefficients in this study were 0.93, respectively and KMO test value was 0.927, which showed good reliability and validity.

SECONDARY OUTCOMES:
Illness Perception | From enrollment through study completion, an average of 6 months
  The investigators administered the Brief Illness Perception Questionnaire (BIPQ) to assess the dyads' cognitive and emotional reactions to illness. The scale has 9 items, with items 1-5 assessing cognition, items 6 and 8 assessing emotional status, item 7 assessing comprehension, and item 9 being an open-ended question about causality of the cause of the illness. Each item is scored on a scale of 0 to 10, and the total score ranges from 0 to 80, with higher scores indicating more negative perceptions of the illness. Cronbach's alpha coefficient in this study was 0.77.
mindfulness | From enrollment through study completion, an average of 6 months
  The investigators used the Mindful Attention Awareness Scale (MAAS) to assess the dyads' mindfulness tendencies. The scale consists of 15 items and each item is assigned a score from 1 to 6, with the scale ranging from "almost always" to "almost never", with higher scores indicating higher levels of awareness and attention to the present moment. Cronbach's alpha coefficient in this study was 0.92.
self-compassion | From enrollment through study completion, an average of 6 months
  The dyadic self-compassion was assessed using the Self-compassion Scale (SCS), which includes six dimensions of self-kindness, self-criticism, common humanity, loneliness, stillness, and over-indulgence, with a total of 26 items, has a high re-test reliability (r=0.93) and internal consistency reliability (α=0.92). Cronbach's α coefficient in this study was 0.88.
dyadic coping | From enrollment through study completion, an average of 6 months
  The Dyadic Coping Inventory (DCI)(32) was used to evaluate the coping ability of dyads. The Chinese version has a total of 37 items, including six dimensions: stress communication, support, negativity, empowerment coping, cooperation, and evaluation. A 5-point Likert scale was used, with higher scores indicating higher levels of positive dyadic coping, and the negative supportive coping items (items 7, 10, 11, 15, 22, 25, 26, 27) were reverse scored, with higher scores indicating higher levels of negative dyadic coping. A total score below 111 is considered low, a total score between 111 and 145 is considered moderate, and a total score above 145 is considered high. Cronbach's alpha coefficients in this study were 0.93.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya School of Nursing, Changsha, China

REFERENCES:
- [Derived] Li J, Li C, Zou J, Cheng FQ, Peng L, Deng LH, Wu PP, Gao SY, Xiong ZY, Zuo Y, Luo Y, Rao XH, Yuan B, Chen OY, Zhang JP. Prevalence and influencing factors of the dyadic psychological stress among patients with lung cancer and their family caregivers: a cross-sectional study. BMC Nurs. 2025 Jan 6;24(1):13. doi: 10.1186/s12912-024-02635-z. PMID 39762831